CLINICAL TRIAL: NCT03574142
Title: A Phase I, Open-label Study to Evaluate the Pharmacokinetics of Single and Multiple Doses of Epanova® in Chinese Healthy Subjects Living in China
Brief Title: A Ph 1 Study of Epanova® in Healthy Chineses
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5881C00001
Record Dates: First submitted 2018-05-04; First posted 2018-06-29 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Healthy Subjects
Keywords: Pharmacokinetics; Safety; Tolerability; Epanova; Omega-3 carboxylic acids; Chinese

STUDY DESIGN:
Intervention Model Description: Single group
Masking Description: Open-label Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epanova (Experimental): Epanova® capsule, per oral
  Interventions: Drug: Epanova

INTERVENTIONS:
Drug: Epanova — A single dose of Epanova 4 g will be administered as 4 capsules (each containing 1 g of Epanova) followed by a 72-hour washout period in Chinese healthy subjects. Subsequently, multiple doses of Epanova 4 g will be administered once daily for 14 consecutive days.
  Other Names: Omega-3 carboxylic acids

SUMMARY:
The purpose of this study is to explore the safety, tolerability, and PK of single and multiple doses of Epanova in healthy male and female Chinese subjects and to allow comparison of these parameters with the Western population studied to date.

DETAILED DESCRIPTION:
This is a single centre, open-label, single- and multiple-dose, PK study in Chinese healthy subjects. Approximately 14 subjects will receive a single oral dose of Epanova 4 g followed by a 72-hour washout period, and then receive Epanova 4 g orally once daily for 14 consecutive days. Subjects will undergo screening evaluations to determine eligibility within 4 weeks (28 days) prior to the first dose of investigational product (IP). Subjects will be admitted to the clinical pharmacology unit approximately 48 hours prior to the first dosing (Day -2) and will stay at the unit until at least 72 hours (Day 20) after their last dose of IP (Day 17). Blood samples will be collected for PK analyses. Subjects will be monitored closely for adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to give written informed consent by signing an IRB-approved Informed Consent Form (ICF) prior to admission to this study and follow the restrictions and procedures outlined for the study.
2. Healthy adult males or females as determined by medical history, physical examination, and laboratory tests. Subjects are to be native Chinese, 18 to 45 years of age (inclusive) at the time of consent.
3. Body mass index (BMI) ≥19 and ≤26 kg/m2 and weigh at least 50 kg.
4. Medically healthy subjects with clinically insignificant screening results (eg, laboratory profiles, medical histories, electrocardiograms [ECGs], physical examination). Haemoglobin must be greater than the lower limit of normal. A 12-lead ECG with QTcF >340 msec and <450 msec.
5. Acceptable supine blood pressure (BP) and heart rate as determined by the investigator (systolic BP ≤140 mm Hg, and diastolic BP ≤90 mm Hg).
6. For women of childbearing potential (have not had tubal ligation, hysterectomy or surgical procedure for sterilisation), the results from a serum pregnancy test at screening and at Day -2 must be within the normal range. The subject must also agree to use an acceptable method of contraception throughout the trial. Women with an intact uterus are deemed postmenopausal if they are at least age 45, have had cessation of menses for at least 1 year, and have not taken hormones or oral contraceptives (including oestrogen or hormone replacement therapy) during the past 12 months.

Key Exclusion Criteria

1. Past history of psychological or physical disorder.
2. An individual who has abnormal laboratory values or an inappropriate current or past medical history for participation based on the PI's decision.
3. Has a history or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease.
4. Has a positive urine drug/alcohol breath testing at the screening visit or on Day -2.
5. Habitual users of drug(s) of abuse.
6. Has tested positive for human immunodeficiency virus (HIV), hepatitis B (including surface antigen [HbsAg] positive healthy carrier), hepatitis C antibodies (HCV), or syphilis.
7. Has used fish oil, other EPA and/or DHA containing supplements within 60 days of admission to the clinic.
8. Has a known sensitivity or allergy to soybeans, fish, and/or shellfish.
9. Has had a history of hypersensitivity or idiosyncratic reaction to compounds related to Epanova.
10. Pregnant or lactating women.
11. Those who have difficulty with blood sampling via a peripheral vein.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
1. Plasma concentrations versus time profile of EPA and DHA | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects
2. Observed maximum plasma concentration (Cmax) | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects
3. Time to reach maximum plasma concentration (tmax) | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects
4. Terminal half-life | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects
5. Area under the plasma concentration-time curve from time zero to time of last quantifiable analyte concentration (AUC0-t)), from time zero to 24 hours (AUC0-24h), and from time zero extrapolated to infinity (AUC) | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects
6. Apparent clearance for parent drug estimated as dose divided by AUC (CL/F) | Blood sample will be collected on Day-1, Day1(-1h, -5min Pre-dose and 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose),Day2,3,4,7,11,14,16,and Day17 (-5min Pre-dose, 1h, 2h, 3h, 4h, 5h, 6h, 7.5h, 9h, 12h, 16h Post-dose), Day18,19 and Day20
  To evaluate the PK of single and multiple oral doses of Epanova in Chinese healthy subjects

SECONDARY OUTCOMES:
Number of subjects with adverse events. | Adverse event will be collected from Visit 4(Day1) to Visit 23 (Day20).
  Following categories will be collected and analyzed: any adverse event (AE), any AE causally related to investigational product (IP), serious adverse events (SAEs), SAEs causally related to IP, AEs with outcome of death, AEs leading to discontinuation of IP, and other significant AEs.
Safety as determined by evaluation of blood pressure in mmHg | Blood presure will be collected from Visit1(any day between Day-28 to Day-2) to Visit23(Day20).
  Measurement of blood pressure (systolic and diastolic in mmHg)
Safety as determined by evaluation of heart beat in beats per minute | Heart beat will be collected from Visit1(any day between Day-28 to Day-2) to Visit23(Day20).
  Measurement of heart beat in beats per minute
Safety as determined by evaluation of body temperature in degree Celsius | Body temperature will be collected from Visit1(any day between Day-28 to Day-2) to Visit23(Day20).
  Measurement of body temperature in degree Celsius
Safety as determined by evaluation of respiratory rate in breaths per minute | Respiratory rate will be collected from Visit1(any day between Day-28 to Day-2) to Visit23(Day20).
  Measurement of respiratory rate in breaths per minute
Safety as determined by analysis of electrocardiograms | Electrocardiograms will be collected at Visit1(any day between Day-28 to Day-2), Visit3(Day-1) and V23(Day20).
  Analysis of 12-lead electorcardiograms
Safety as determined by abnormality in haematology | Blood samples will be collected at Visit1(any day between Day-28 to Day-2), Visit2 (Day -2) and Visit23(Day20).
  Measurement of red blood cell count, white blood cell count, haemoglobin and platelets
Safety as determined by abnormality in clinical chemistry | Blood samples will be collected at Visit1(any day between Day-28 to Day-2), Visit2 (Day -2) and Visit23(Day20).
  Measurement of kidney function (e.g.urea ,creatinine, Uric acid), liver function(ALP, ALT, AST, albumin, total bilirubin, direct bilirubin), lipid profile(total cholesterol, triglycerides), potassium and hs-CRP
Safety as determined by abnormality in urinalysis | Urine samples will be collected at Visit1(any day between Day-28 to Day-2), Visit2 (Day -2) and Visit23(Day20).
  Measurement of leucocyte, red blood cells, protein and microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Yang Lin, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Research Site, Beijing, China

IPD SHARING:
Plan to Share IPD: No